CLINICAL TRIAL: NCT01197560
Title: A Phase 2/3, Multicenter, Randomized, Open-label Study to Compare the Efficacy and Safety of Lenalidomide (Revlimid ®) Versus Investigator's Choice in Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma
Brief Title: Study of Lenalidomide to Evaluate Safety and Effectiveness in Patients With Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-DLC-001
Record Dates: First submitted 2010-07-29; First posted 2010-09-09 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Diffuse Large B-Cell Lymphoma; Non Hodgkin's Lymphoma; relapsed; refractory; relapsed/refractory; DLBCL; Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Recurrence | interventions — Lenalidomide; Gemcitabine; Oxaliplatin; Rituximab; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lenalidomide (Experimental): Lenalidomide 25 mg capsules by mouth on days 1-21 of each 28 day cycle. For patients with Creatinine Clearance ≥ 30 mL/min but < 60 mL/min, lenalidomide 10 mg (max escalation is 15 mg).
  Interventions: Drug: Lenalidomide
- Investigators Choice (Active Comparator): One of the following:
  Gemcitabine, Oxaliplatin, Rituximab, or Etoposide
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Rituximab; Drug: Etoposide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide 25 mg orally for 21/28 days until Diffuse Large B-Cell Lymphoma (DLBCL) progressive disease. For patients with Creatinine Clearance ≥ 30 mL/min but < 60 mL/min, lenalidomide 10 mg (max escalation is 15 mg).
  Arms: Lenalidomide
Drug: Gemcitabine — Suggested starting doses and regimens for Gemcitabine is 1,250 mg/m^2 intravenous (IV) administration on days 1, 8, 15 every 28 days for 6 Cycles or 1,000 mg/m^2 IV days 1 and 15 every 28 days for 6 Cycles
  Arms: Investigators Choice
Drug: Oxaliplatin — Suggested starting dose and regimen for Oxaliplatin is 100 mg/m^2 IV day 1 for 21 days for 6 Cycles
  Arms: Investigators Choice
Drug: Rituximab — Suggested starting dose for Rituximab is 375 mg/m^2 IV days 1, 8, 15, 22 during Cycle 1, and if stable disease at Week 12, also on Day 1 of Cycles 4, 6, 8, and 10 (CD20+ patients only)
  Arms: Investigators Choice
Drug: Etoposide — Suggested starting doses for Etoposide are:
  100 mg/m^2 IV days 1-5 every 28 days for 6 Cycles, or 100 mg/m^2 IV days 1-3 every 28 days for 6 Cycles, or 50 mg/m^2 oral days 1-21 every 28 days for 6 Cycles, or 50 mg/m^2 oral days 1-14 every 28 days for 6 Cycles, or 50 mg/m^2 oral days 1-10 every 28 days for 6 Cycles
  Arms: Investigators Choice

SUMMARY:
The purpose of this study is to compare lenalidomide to a control drug and see which one delays Diffuse Large B-Cell Lymphoma (DLBCL) disease progression longer.

DETAILED DESCRIPTION:
This research study is for patients who have been diagnosed with Diffuse Large B-cell Lymphoma (DLBCL) that did not respond to (refractory) or that has come back after chemotherapy treatment (relapsed). Lymphoma is a cancer of a type of blood cell called lymphocytes. DLBCL is just one type of lymphoma. Within DLBCL there are two different subtypes called Germinal Center B-cell (GCB) and non-GCB which can be determined by cell surface marker tests or by gene expression tests. Scientists can look at cells and genes in the laboratory and see that the two kinds are different, but they don't know yet what the difference means. To patients and doctors these two kinds seem the same. Right now doctors don't usually do tests to find out which kind a patient has because the treatment is the same for both.

This study will have two stages, 1 and 2. The main purpose of Stage 1 is to separate patients by subtype and then test whether patients taking lenalidomide or any one of four other drugs have a better response. It is possible that lenalidomide will work better than one of the other drugs in zero, one, or both subtypes. Stage 2 will further test only the subtype(s) from Stage 1 that showed a good response to lenalidomide. The main purpose of Stage 2 is to test how long patients are disease free on lenalidomide compared to one of the four other drugs.

On 29 January 2013 the enrolment goal for the Stage 1 portion of the study was met and enrollment was stopped. The final analysis for Stage 1 was performed as of the 04 Jul 2013 data cutoff date. According to the Stage 1 results as assessed by the independent response adjudication committee (IRAC), neither subtype met the pre specified requirement to be further studied in Stage 2. Additionally, a suitable assay for the selection of participants for the Stage 2 study was not available. Therefore, on 6 January 2014, Celgene decided to not open Stage 2.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven Diffuse Large B-Cell Lymphoma (DLBCL).
* Relapsed or refractory to combination chemotherapy for DLBCL that contains rituximab and an anthracycline, and one additional combination chemotherapy or stem cell transplant.
* Measurable DLBCL disease by computed tomograph (CT) / magnetic resonance imagining (MRI).
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2.

Exclusion Criteria:

* Diagnosis of lymphoma histologies other than DLBCL.
* History of malignancies, other than DLBCL, unless the patient has been disease free for 3 years or more.
* Eligible for autologous stem cell transplant.
* Known seropositive for, or history of, active human immunodeficiency virus (HIV) hepatitis B virus (HBV), hepatitis C virus (HCV)
* Neuropathy grade 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2010-09-02 (Actual); Primary Completion 2013-07-04 (Actual); Study Completion 2018-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Kilcoyne, MD, Study Director — Celgene Corporation
Locations (57):
- United States (13):
  - Providence St Joseph Medical Center/Cancer Center, Burbank, California
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - University of Michigan, Comprehensive Cancer Center, Ann Arbor, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Washington University Siteman Cancer Center, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Houston, Houston, Texas
- Australia (3):
  - Royal Adelaide Hospital, Adelaide
  - Royal Brisbaine and Womens Hospital, Herston
  - Princess Alexandra Hospital, Woolloongabba
- Austria (3):
  - Innsbruck University Hospital, Innsbruck
  - Universitätsklinikum Salzburg, Salzburg
  - Medical University of Vienna, Vienna
- Czechia (2):
  - University Hospital Hradec Kralove, Hradec Králové
  - Charles University, Prague
- France (11):
  - ICH CHU Brest- C.H.U. MORAVAN, Brest
  - CHU de Grenoble-Hopital Albert Michallon, Grenoble
  - Chd -Vendee, La Roche-sur-Yon
  - Centre Hospitalier Lyon Sud, Lyon
  - Institute Paoli-Calmette, Marsielle
  - Hotel Dieu, Nantes
  - Hôpital Saint Jean, Perpignan
  - CHRU-Hopital du Haut -Leveque, Pessac
  - CHU de Rennes Hopital de Pontchaillou, Rennes
  - University Hospital OF Toulouse Purpan, Toulouse
  - Hopital de Brabois Adultes, Vandœuvre-lès-Nancy
- Italy (9):
  - Istituto di Ematologica Istituto di Ematologica " L.e. A. Seragnoli' Azienda Ospedaliera Universitaria Policlinico, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Clinica Ematologica, A.O.U. San Martino di Genova, Genova
  - IEO istituto Europeo di Oncologia, Miano
  - Universita Federico II di Napoli Nuovo Policlinico, Napoli
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Irccs/Crob, Rionero in Vulture (PZ)
  - Policlinico Tor Vergata (Universta Tor Vergata), Roma
  - Azienda Ospedaliera di Perugai Ospedale S. Maria della Miseri, Terni
- Spain (6):
  - Hospital Universitari Vll D' Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Costa Del Sol, Marbella
  - CH de Orense, Ourense
  - Complejo Hospitalario de Navarra, Pamplona
  - Hosptial Clinico Universitario de Salamanca, Salamanca
- Sweden (2):
  - Onkologiska kliniken, Umeå
  - Akademiska Sjukhuset, Uppsala
- United Kingdom (8):
  - Royal Bournemouth Hospital Haematology, Bournemouth
  - Royal Devon and Exeter Hospital Haematology Department, Exeter
  - St. James Institute of Oncology, Leeds
  - Royal Mardsen Hospital - Fulham (Satellite Site), London
  - The Christie Foundation Trust, I'st Floor, Haemotology Oncology Outpatients, Lymphoma Team, Manchester
  - Derrford Hospital, Plymouth
  - Southhampton University Hospital NHS Trust, Southhampton
  - Royal Mardsen NHS Foundation Trust, Sutton

REFERENCES:
- [Result] Czuczman MS, Trneny M, Davies A, Rule S, Linton KM, Wagner-Johnston N, Gascoyne RD, Slack GW, Brousset P, Eberhard DA, Hernandez-Ilizaliturri FJ, Salles G, Witzig TE, Zinzani PL, Wright GW, Staudt LM, Yang Y, Williams PM, Lih CJ, Russo J, Thakurta A, Hagner P, Fustier P, Song D, Lewis ID. A Phase 2/3 Multicenter, Randomized, Open-Label Study to Compare the Efficacy and Safety of Lenalidomide Versus Investigator's Choice in Patients with Relapsed or Refractory Diffuse Large B-Cell Lymphoma. Clin Cancer Res. 2017 Aug 1;23(15):4127-4137. doi: 10.1158/1078-0432.CCR-16-2818. Epub 2017 Apr 5. PMID 28381416
- [Derived] Hernandez-Ilizaliturri FJ, Deeb G, Zinzani PL, Pileri SA, Malik F, Macon WR, Goy A, Witzig TE, Czuczman MS. Higher response to lenalidomide in relapsed/refractory diffuse large B-cell lymphoma in nongerminal center B-cell-like than in germinal center B-cell-like phenotype. Cancer. 2011 Nov 15;117(22):5058-66. doi: 10.1002/cncr.26135. Epub 2011 Apr 14. PMID 21495023

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening and enrollment occurred at 43 sites, including 10 in the United States, 9 in France, 7 in the United Kingdom; 4 in Spain, 4 in Italy, 3 each in Austria and Australia, 2 in the Czech Republic, and 1 in Sweden.
Pre-assignment Details: Participants were stratified into Germinal center B-cell (GCB) or non-GCB subtypes and randomized 1:1 to receive lenalidomide or investigator's choice treatment (one of the single-agent reference therapies [gemcitabine, rituximab, etoposide, or oxaliplatin)
Groups:
- Lenalidomide: Participants received lenalidomide 25 mg orally once daily for 21 days in each 28-day cycle until progressive disease. For participants with creatinine clearance ≥ 30 mL/min but < 60 mL/min, lenalidomide 10 mg once daily for 21 days for 2 cycles. After Cycle 2 the dose may have been increased to a maximum of 15 mg lenalidomide once daily for 21 days in each 28-day cycle. Treatment was continued until disease progression, unacceptable toxicity, or voluntary withdrawal.
- Investigators Choice (Control Arm): Participants received a single agent reference therapy (either gemcitabine, oxaliplatin, rituximab or etoposide) based on published data for up to 6 cycles or until disease progression, unacceptable toxicity or withdrawal. Participants with documented progressive disease had the option to receive crossover lenalidomide at the same dosage as participants randomized to lenalidomide.
Period: Overall Study
Arm/Group | Lenalidomide | Investigators Choice (Control Arm)
Started | 54 (This is the intent to treat population) | 57 (This is the intent to treat population)
Received ≥ One Dose Study Drug | 54 | 55
Lenalidomide Crossover | 0 | 29
Discontinued Treatment After ≥ 6 Cycles | 14 | 0
Completed (Completed indicates the participates who completed core treatment.) | 0 | 4
Not Completed | 54 | 53
Not completed — Adverse Event | 6 | 8
Not completed — Death | 3 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Disease progression | 40 | 35
Not completed — Miscellaneous | 4 | 3
Not completed — Missing | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat (mITT) = all study participants randomized with a diffuse large B-cell lymphoma (DLBCL) diagnosis and germinal center B-cell (GCB)/non-germinal center B (non-GCB) subtype confirmed by central pathology, and who received at least one dose of study drug (lenalidomide or Investigator's choice). Nine participants were excluded.
Groups:
- Investigators Choice (IC): Participants received a single agent reference therapy (either gemcitabine, oxaliplatin, rituximab or etoposide) based on published data for up to 6 cycles or until disease progression, unacceptable toxicity or withdrawal. Gemcitabine 1,250 mg/m^2 Intravenous (IV) days 1, 8, 15 every 28 days for 6 Cycles or 1,000 mg/m^2 IV days 1 and 15 in each 28- day cycle for 6 Cycles Oxaliplatin 100 mg/m^2 IV day 1 in each 21-day cycle for 6 Cycles Rituximab is 375 mg/m^2 IV days 1, 8, 15, 22 during Cycle 1, and if stable disease at Week 12, also on Day 1 of Cycles 4, 6, 8, and 10 (CD20+ patients only) Etoposide doses: 100 mg/m^2 IV days 1-5 in each 28-day cycle for 6 Cycles, or 100 mg/m^2 IV days 1-3 in each 28-day cycle for 6 Cycles, or 50 mg/m^2 oral days 1-21 in each 28-day cycle for 6 Cycles, or 50 mg/m^2 oral days 1-14 in each 28-day cycle for 6 Cycles, or 50 mg/m^2 oral days 1-10 in each 28-day cycle for 6 Cycles
- Total: Total of all reporting groups
Arm/Group | Lenalidomide | Investigators Choice (IC) | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (13.43) | 62.8 (13.94) | 63.75 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 30 | 31 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Black/African American | 0 | 1 | 1
  White | 38 | 36 | 74
  Missing | 9 | 11 | 20
  Other (Unspecified) | 3 | 2 | 5
Eastern Cooperative Oncology Performance Status (ECOG)] [Count of Participants; unit: Participants] — ECOG performance status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the subject and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  Participants
    0 = (Fully Active) | 18 | 15 | 33
    1 (Restrictive but Ambulatory) | 24 | 28 | 52
    2 (Ambulatory but Unable to Work) | 7 | 8 | 15
    3 (Limited Self-Care) | 0 | 0 | 0
    4 (Completely Disabled) | 1 | 0 | 1
    Missing | 1 | 0 | 1
Creatinine Clearance (CrCl) [Count of Participants; unit: Participants] — Creatinine is a waste product from the normal breakdown of muscle tissue. As creatinine is produced, it's filtered through the kidneys and excreted in urine. Doctors measure the blood creatinine level as a test of kidney function. Participants with a CrCl (as calculated by the Cockcroft-Gault formula, utilizing actual body weight or ideal body weight, whichever was less) of ≥ 60 mL/min received a starting dose of 25 mg lenalidomide once daily. Participants with moderate renal insufficiency (ie, CrCl ≥ 30 mL/min but < 60 mL/min) received a starting dose of 10 mg lenalidomide once daily.
  Participants
    ≥ 60 mL/min | 32 | 43 | 75
    ≥ 30 but < 60 mL/min | 18 | 7 | 25
    Missing | 1 | 1 | 2
Disease Stage of DLBCL at Enrollment [Count of Participants; unit: Participants] — The criteria for Clinical Stage (Ann Arbor staging) are as below: I: involvement of a single nodal region. II: involvement of 2 or more lymph node regions on the same side of the diaphragm. III: involvement of lymph node regions on both sides of the diaphragm. IV: disseminated involvement of 1 or more extra-lymphatic sites with or without associated lymph node involvement. A or B: the absence of constitutional (B-type) symptoms is denoted by adding an "A" to the stage; the presence is denoted by adding a "B" to the stage.
  Participants
    IA | 1 | 3 | 4
    IB | 1 | 0 | 1
    IIA | 8 | 7 | 15
    IIB | 3 | 1 | 4
    IIIA | 13 | 13 | 26
    IIIB | 2 | 4 | 6
    IVA | 17 | 14 | 31
    IVB | 6 | 9 | 15
Diffuse Large B-Cell Lymphoma (DLBCL) Subtypes - Germinal Center B-Cell (GCB) and non-GCB [Count of Participants; unit: Participants] — DLBCL is comprised of different pathophysiological subtypes that influence patient prognosis and response to treatment. Based on immunohistochemistry (IHC), DLBCL can be classified into germinal center B-cell (GCB) and non-GCB subtypes. Patients with non-GCB have a worse prognosis compared with the GCB subtype Population: The Modified Intent to Treat (mITT ) population was defined as all participants randomized who had a DLBCL diagnosis and either Germinal Center B-cell subtype or non-GCB subtype confirmed by central pathology, and who received at least one dose of study drug (lenalidomide or investigator's choice).
  Participants
    Germinal Center B-Cell Type | 23 | 25 | 48
    Non-Germinal Center B-Cell Type | 28 | 26 | 54

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Percentage of Participants With an Overall Response According to the International Working Group (IWG) Response Criteria for Non Hodgkin's Lymphoma (NHL), Cheson 1999 and Evaluated by the Independent Response Adjudication Committee (IRAC)
Description: An overall response is a complete response (CR), unconfirmed complete response (CRu) or partial response (PR) and was evaluated by the IRAC. A CR = complete disappearance of disease and related symptoms. Lymph nodes and nodal masses regressed on computed tomography to normal size (≤ 1.5 cm in their greatest transverse diameter for nodes > 1.5 cm prior to therapy and ≤ 1.0 cm in their short axis for nodes 1.1-1.5 cm in their long axis and > 1.0 cm in their short axis prior to therapy). Spleen and/or liver not palpable on exam, normal size by imaging, and absence of nodules related to lymphoma. If bone marrow was involved prior to therapy, infiltrate must have cleared on repeat biopsy. PR = ≥ 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses. No increase in other nodes, liver, or spleen. Splenic and hepatic nodules regressed by ≥ 50% in their SPD or for single nodules, in the greatest transverse diameter;no new disease.
Time Frame: From the date of randomization to the data cut-off of 4 July 2013; when all patients reached the scheduled 16-week assessment or had progressed/died before the scheduled 16-week assessment); the median study duration was 27.0 and 19.7 weeks, respectively.
Population: The Modified Intent to Treat (mITT) population was defined as all participants randomized who had a diffuse large B-cell lymphoma (DLBCL) diagnosis and either germinal center B-cell subtype (GCB) or non-GCB subtype confirmed by central pathology, and who received at least one dose of study drug (lenalidomide or investigator's choice).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide | Investigators Choice (IC)
Number analyzed (Participants) | 51 | 51
percentage of participants
  ORR for All Participants | 27.5 [15.9 to 41.7] | 11.8 [4.4 to 23.9]
  GCB Subtype: number analyzed (Participants) | 23 | 25
  GCB Subtype | 26.1 [10.2 to 48.4] | 12.0 [2.5 to 31.2]
  Non-GCB: number analyzed (Participants) | 28 | 26
  Non-GCB | 28.6 [13.2 to 48.7] | 11.5 [2.4 to 30.2]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice (IC); Pertains to all participants; row 1; Test type: Superiority; p = 0.079, Fisher Exact
Statistical Analysis 2: Comparison: Investigators Choice (IC); Pertains to GCB Subtype; row 2; Test type: Superiority; p = 0.279, Fisher Exact
Statistical Analysis 3: Comparison: Investigators Choice (IC); Pertains to non-GCB Sub-type; row 3; Test type: Superiority; p = 0.179, Fisher Exact

2. Primary Outcome: Stage 1: Percentage of Participants With an Overall Response According to the IWG Response Criteria Based on the Investigators Assessment at the Final Data Cut During the Core Treatment Phase
Description: Response was defined as having a CR, CRu or PR, based on IWG 1999 Response Criteria for NHL as evaluated by the investigators. CR = complete disappearance of disease and disease related symptoms. All lymph nodes and nodal masses regressed on computed tomography to normal size (≤ 1.5 cm in their greatest transverse diameter for nodes > 1.5 cm prior to therapy and ≤ 1.0 cm in their short axis for nodes 1.1-1.5 cm in their long axis and > 1.0 cm in their short axis prior to therapy). Spleen and/or liver not palpable on physical exam, normal size by imaging, and absence of nodules related to lymphoma. If BM was involved prior to therapy, infiltrate must have cleared on repeat biopsy. PR = ≥ 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses. No increase in the other nodes, liver, or spleen. Splenic and hepatic nodules regressed by ≥ 50% in their SPD or, for single nodules, in the greatest transverse diameter. No new disease.
Time Frame: From the date of randomization to the final data cut-off date of 18 May 2018; median study duration was 27.0 and 19.7 weeks, respectively.
Population: mITT was defined as all participants randomized who had a DLBCL diagnosis confirmed by central pathology, had either GCB or non-GCB subtype and received at least one dose of study drug or investigators choice regimen.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenalidomide | Investigators Choice (IC)
Number analyzed (Participants) | 51 | 51
Percentage of participants | 29.4 [17.5 to 43.8] | 13.7 [5.7 to 26.3]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice (IC); Pertains to all participants; Test type: Superiority; p = 0.091, Fisher Exact

3. Other Pre Specified Outcome: Stage 1: Percentage of Participants With a Durable Overall Response (dORR) According to the IWG Response Criteria as Assessed by the Investigators at the Final Data Cut During the Core Treatment Phase
Description: Durable overall response rate was defined as the percentage of participants who maintained a response for at least 16 weeks after initial response.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide | Investigators Choice (Control Arm)
Number analyzed (Participants) | 51 | 51
percentage of participants | 23.5 [12.8 to 37.5] | 9.8 [3.3 to 21.4]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice (Control Arm); Test type: Superiority; p = 0.109, Fisher Exact

4. Other Pre Specified Outcome: Stage 1: Percentage of Participants With a Complete Response According to the IWG Response Criteria as Assessed by the Investigators at the Final Data Cut During the Core Treatment Phase
Description: A complete response was defined as participants with a complete response (CR), or unconfirmed complete response (CRu) based on IWG 1999 Response Criteria for NHL as assessed by the investigator. A CR is a complete disappearance of all disease with the exception of nodes. No new lesions. Previously enlarged organs must have regressed and not be palpable. Bone marrow must be negative if positive at baseline. Normalization of markers. CR Unconfirmed (CRu) does not qualify for CR above, due to a residual nodal mass or an indeterminate BM.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide | Investigators Choice (IC)
Number analyzed (Participants) | 51 | 51
percentage of participants | 13.7 [5.7 to 26.3] | 3.9 [0.5 to 13.5]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice (IC); Pertains to all participants; row 1; Test type: Superiority; p = 0.160, Fisher Exact

5. Other Pre Specified Outcome: Stage 1: Kaplan Meier Estimates of Duration of Overall Response (DoR) as Assessed by the Investigators at the Final Data Cut During the Core Treatment Phase
Description: Duration of overall response was calculated as the time of initial response (CR+CRu+PR) until documented disease progression determinted by computerized scan CT scan or MRI or death due to lymphoma, whichever occurred earlier, for participants who responded.
Time Frame: as for outcome 2
Population: For DoR, the population included participants who had an overall response.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Lenalidomide | Investigators Choice (Control Arm)
Number analyzed (Participants) | 15 | 7
Weeks | 64.7 [29.1 to 141.6] | 63.1 [15.3 to 79.4]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice (Control Arm); Test type: Superiority; p = 0.529, Log Rank

6. Other Pre Specified Outcome: Stage 1: Kaplan Meier Estimates of Duration of Complete Response (DoCR) as Assessed by the Investigators at the Final Data Cut During the Core Treatment Phase
Description: Duration of complete response was defined as the time from the first documented complete response (CR + CRu) until the first disease progression or death for participants who had a CR.
Time Frame: as for outcome 2
Population: For DoCR, the population included participants who had a CR.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Lenalidomide | Investigators Choice (Control Arm)
Number analyzed (Participants) | 7 | 2
Weeks | 66.4 [22.1 to NA] — No estimable due to that the estimated upper 97.5% survival curve does not reach 50%. | 179.3 [63.1 to 295.4]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice (Control Arm); Test type: Superiority; p = 0.972, Log Rank

7. Other Pre Specified Outcome: Stage 1: Kaplan Meier Estimates of Progression-Free Survival As Assessed By The Investigators At The Final Data Cut During The Core Treatment Phase
Description: Progression-free survival was defined as the time from randomization to the first documented disease progression or death due to any cause.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Lenalidomide | Investigators Choice (IC)
Number analyzed (Participants) | 51 | 51
Weeks | 9.6 [7.6 to 17.1] | 7.1 [6.0 to 8.3]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice (IC); Test type: Superiority; p = 0.020, Log Rank

8. Other Pre Specified Outcome: Stage 1: Kaplan Meier Estimates of Overall Survival As Assessed by the Investigators at the Final Data Cut During The Core Treatment Phase
Description: Overall survival was defined as time from randomization until death of any cause.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Lenalidomide | Investigators Choice (IC)
Number analyzed (Participants) | 51 | 51
Weeks | 31.0 [16.6 to 43.7] | 24.6 [12.7 to 34.9]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice (IC); Test type: Superiority; p = 0.211, Log Rank

9. Secondary Outcome: Number of Participants With Treatment Emergent Events (TEAEs) in the Overall Treatment Phase by Initial Treatment Assignment
Description: A TEAE was defined as an AE that begins or worsens in intensity of frequency on or after the first dose of study drug through 28 days after last dose of study drug.
  A serious adverse event (SAE) is any:
  * Death;
  * Life-threatening event;
  * Any inpatient hospitalization or prolongation of existing hospitalization;
  * Persistent or significant disability or incapacity;
  * Congenital anomaly or birth defect;
  * Any other important medical event The investigator determined the relationship of an AE to study drug based on the timing of the AE relative to drug administration and whether or not other drugs, therapeutic interventions, or underlying conditions could provide a sufficient explanation for the event.The severity of an AE was evaluated by the investigator according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (Version 4.03) where Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening and Grade 5 = Death
Time Frame: From first dose of study drug to the final data cut-off date of 18 May 2018; median study duration was 27.0 and 19.7 weeks, respectively.
Population: Safety Population included all participants who received at least one dose of lenalidomide or IC regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide | Investigators Choice (IC)
Number analyzed (Participants) | 54 | 55
Participants
  Any TEAEs | 54 | 55
  Any Treatment Related TEAE | 49 | 45
  Any TEAE Grade ≥ 3 | 43 | 53
  Any TEAE Grade ≥ 4 | 29 | 36
  Any TEAE Grade 5 | 9 | 18
  Any TEAE Grade 3 or 4 | 42 | 52
  Any Treatment Related TEAE Grade ≥ 3 | 30 | 39
  Any Treatment Related TEAEs Grade ≥ 4 | 15 | 21
  Any Treatment Related TEAE Grade 5 | 0 | 2
  Any Treatment Related TEAE Grade 3 or 4 | 30 | 39
  Any Serious Adverse Events (SAEs) | 31 | 42
  Any Treated Related SAEs | 14 | 21
  Any AE leading to stopping of study drug | 11 | 17
  Any drug related AE leading to halt of study drug | 5 | 4
  Any AE leading to dose interruption/reduct | 32 | 34
  Any drug related AE leading to interruption/reduct | 27 | 30

10. Secondary Outcome: Stage 2: Overall Response Rate (ORR)
Description: ORR is defined as: Complete Response + Complete Response unconfirmed + Partial Response based on the International Lymphoma Workshop Response Criteria [IWRC] (Cheson 1999).
Time Frame: Approximately 3.5 years
Population: ORR not analyzed; the Stage 1 results as assessed by the independent response adjudication committee (IRAC), demonstrated that neither subtype met the pre-specified requirement to be further studied in Stage 2. Study terminated after Stage 1 completed and before Stage 2 started.
Arm/Group | Lenalidomide | Investigators Choice (Control Arm)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Stage 2: Duration of Response (DoR)
Description: Length of time of overall response (Complete Response + Complete Response unconfirmed + Partial Response) based on the International Lymphoma Workshop Response Criteria [IWRC] (Cheson 1999).
Time Frame: Approximately 3.5 years
Population: DoR not analyzed; the Stage 1 results as assessed by the independent response adjudication committee (IRAC), demonstrated that neither subtype met the pre-specified requirement to be further studied in Stage 2. Study terminated after Stage 1 completed and before Stage 2 started.
Arm/Group | Lenalidomide | Investigators Choice (Control Arm)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Stage 2: Overall Survival (OS)
Description: Overall survival was defined as time from randomization until death of any cause.
Time Frame: Approximately 3.5 years
Population: OS not analyzed; the Stage 1 results as assessed by the independent response adjudication committee (IRAC), demonstrated that neither subtype met the pre-specified requirement to be further studied in Stage 2. Study terminated after Stage 1 completed and before Stage 2 started.
Arm/Group | Lenalidomide | Investigators Choice (Control Arm)
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Stage 2: Progression-Free Survival
Description: Number of participants who survive without progressing based on the International Working Group Response Criteria [IWG].
Time Frame: Approximately 3.5 years
Population: PFS not analyzed; the Stage 1 results as assessed by the independent response adjudication committee (IRAC), demonstrated that neither subtype met the pre-specified requirement to be further studied in Stage 2. Study terminated after Stage 1 completed and before Stage 2 started.
Arm/Group | Lenalidomide | Investigators Choice (IC)
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Stage 2: Duration of Complete Response
Description: Length of time of complete response (Complete Response + Complete Response unconfirmed) based on the International Lymphoma Workshop Response Criteria [IWRC] (Cheson 1999).
Time Frame: Approximately 3.5 years
Population: Duration of CR was not analyzed; the Stage 1 results as assessed by the independent response adjudication committee (IRAC), demonstrated that neither subtype met the pre-specified requirement to be further studied in Stage 2. Study terminated after Stage 1 completed and before Stage 2 started.
Arm/Group | Lenalidomide | Investigators Choice (Control Arm)
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Stage 2: Overall Response Rate for With a Duration of Response Lasting ≥ 16 Weeks
Description: Complete Response + Complete Response unconfirmed + Partial Response for participants with a duration of response lasting ≥ 16 weeks based on the International Lymphoma Workshop Response Criteria [IWRC] (Cheson 1999).
Time Frame: Approximately 3.5 years
Population: Overall Response Rate for with a Duration of Response Lasting ≥ 16 weeks was not analyzed: the Stage 1 results as assessed by the IRAC, demonstrated that neither subtype met the pre-specified requirement to be further studied in Stage 2. Study terminated after Stage 1 completed and before Stage 2 started.
Arm/Group | Lenalidomide | Investigators Choice (Control Arm)
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Stage 2: Time to Progression
Description: Length of time until disease progression occurs
Time Frame: Approximately 3.5 years
Population: Time to progression was not analyzed; the Stage 1 results as assessed by the IRAC, demonstrated that neither subtype met the pre-specified requirement to be further studied in Stage 2. Study terminated after Stage 1 completed and before Stage 2 started.
Arm/Group | Lenalidomide | Investigators Choice (Control Arm)
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Stage 2: Health Related Quality of Life Questionnaires
Description: Quality of Life based on the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 and the EQ-5D assessments
Time Frame: Approximately 3.5 years
Population: Health Related Quality of Life Instruments were not analyzed; the Stage 1 results as assessed by the IRAC, demonstrated that neither subtype met the pre-specified requirement to be further studied in Stage 2. Study terminated after Stage 1 completed and before Stage 2 started.
Arm/Group | Lenalidomide | Investigators Choice (IC)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug to the final data cut-off date of 18 May 2018; the median study duration of 27.0 and 19.7 weeks, respectively.
Description: The AEs were based on the overall treatment phase that includes both core treatment phase and crossover phase. Two participants in the investigator choice arm elected to discontinue before cycle 1; secondary primary malignancies were monitored up to final database lock of 18 May 2018
Groups:
- Investigator's Choice: Investigator's Choice
Arm/Group | Lenalidomide | Investigator's Choice
All-Cause Mortality (participants affected / at risk) | 48/54 | 51/55
Serious Adverse Events (participants affected / at risk) | 31/54 | 42/55
Other Adverse Events (participants affected / at risk) | 53/54 | 52/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=54) | Investigator's Choice (N=55)
ANAEMIA (Blood and lymphatic system disorders) | 4 | 3
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 0 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 4 | 2
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 3
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 1
DUODENAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0
ILEUS (Gastrointestinal disorders) | 1 | 1
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 | 0
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 0 | 3
ASTHENIA (General disorders) | 0 | 2
DEATH (General disorders) | 1 | 0
FATIGUE (General disorders) | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 2
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 1
PERFORMANCE STATUS DECREASED (General disorders) | 0 | 1
PYREXIA (General disorders) | 2 | 2
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 4
DIARRHOEA INFECTIOUS (Infections and infestations) | 0 | 1
GASTROENTERITIS (Infections and infestations) | 1 | 1
INFECTION (Infections and infestations) | 1 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
LUNG ABSCESS (Infections and infestations) | 0 | 1
LUNG INFECTION (Infections and infestations) | 1 | 1
LYMPH NODE ABSCESS (Infections and infestations) | 0 | 1
NEUTROPENIC SEPSIS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 3 | 3
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 1 | 2
SEPTIC SHOCK (Infections and infestations) | 1 | 2
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 | 1
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 2 | 0
WOUND INFECTION (Infections and infestations) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 0 | 1
BLOOD CREATININE INCREASED (Investigations) | 0 | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 3
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 2
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 10
GASTROINTESTINAL TRACT ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RECTOSIGMOID CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
TUMOUR FLARE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CAUDA EQUINA SYNDROME (Nervous system disorders) | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 0 | 1
NERVE ROOT COMPRESSION (Nervous system disorders) | 0 | 1
SEIZURE (Nervous system disorders) | 1 | 1
ANXIETY (Psychiatric disorders) | 0 | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 2
HYDRONEPHROSIS (Renal and urinary disorders) | 1 | 0
NEPHROTIC SYNDROME (Renal and urinary disorders) | 1 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 1
LARYNGEAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PHARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 1
STRIDOR (Respiratory, thoracic and mediastinal disorders) | 1 | 0
FUNGATING WOUND (Skin and subcutaneous tissue disorders) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
EMBOLISM (Vascular disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=54) | Investigator's Choice (N=55)
ANAEMIA (Blood and lymphatic system disorders) | 17 | 31
LEUKOPENIA (Blood and lymphatic system disorders) | 3 | 8
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 | 5
NEUTROPENIA (Blood and lymphatic system disorders) | 23 | 18
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 13 | 17
TACHYCARDIA (Cardiac disorders) | 3 | 1
HYPOACUSIS (Ear and labyrinth disorders) | 0 | 3
VERTIGO (Ear and labyrinth disorders) | 3 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 4 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 10 | 12
CONSTIPATION (Gastrointestinal disorders) | 16 | 16
DIARRHOEA (Gastrointestinal disorders) | 18 | 16
DRY MOUTH (Gastrointestinal disorders) | 7 | 3
DYSPEPSIA (Gastrointestinal disorders) | 3 | 3
NAUSEA (Gastrointestinal disorders) | 10 | 23
STOMATITIS (Gastrointestinal disorders) | 1 | 5
VOMITING (Gastrointestinal disorders) | 9 | 11
ASTHENIA (General disorders) | 10 | 13
CHILLS (General disorders) | 4 | 2
FATIGUE (General disorders) | 19 | 16
NON-CARDIAC CHEST PAIN (General disorders) | 4 | 1
OEDEMA PERIPHERAL (General disorders) | 9 | 10
PYREXIA (General disorders) | 16 | 18
BRONCHITIS (Infections and infestations) | 6 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 6
LUNG INFECTION (Infections and infestations) | 0 | 3
NASOPHARYNGITIS (Infections and infestations) | 3 | 1
PNEUMONIA (Infections and infestations) | 1 | 3
RHINITIS (Infections and infestations) | 3 | 4
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 | 5
URINARY TRACT INFECTION (Infections and infestations) | 3 | 4
DRUG PRESCRIBING ERROR (Injury, poisoning and procedural complications) | 5 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 4
BLOOD CREATININE INCREASED (Investigations) | 2 | 4
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 | 3
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 3
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 7
PLATELET COUNT DECREASED (Investigations) | 0 | 9
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 5
DECREASED APPETITE (Metabolism and nutrition disorders) | 8 | 15
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 | 6
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 6 | 10
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 8
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 4 | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 | 4
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 | 5
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
TUMOUR FLARE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
DIZZINESS (Nervous system disorders) | 3 | 5
DYSGEUSIA (Nervous system disorders) | 2 | 3
HEADACHE (Nervous system disorders) | 3 | 6
HYPOAESTHESIA (Nervous system disorders) | 3 | 1
LETHARGY (Nervous system disorders) | 4 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 | 5
ANXIETY (Psychiatric disorders) | 4 | 5
DEPRESSION (Psychiatric disorders) | 3 | 3
INSOMNIA (Psychiatric disorders) | 3 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 13 | 10
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 | 12
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 3
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 4
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 3 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 3 | 3
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1 | 3
RASH (Skin and subcutaneous tissue disorders) | 9 | 2
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 3 | 1
HYPOTENSION (Vascular disorders) | 3 | 3

LIMITATIONS AND CAVEATS:
On 29 January 2013 the Stage 1 portion of the study was met and enrollment stopped. The Stage 1 results as assessed by the IRAC demonstrated that neither subtype met the prespecified requirement to be further studied in Stage 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.